CLINICAL TRIAL: NCT01471535
Title: HBsAg Loss/Seroconversion in Inactive Chronic Hepatitis B Carriers Treated With Peginterferon Alpha-2a
Brief Title: HBsAg Clearance in Inactive Chronic HBsAg Carriers After Interferon Treated
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of division 4, liver diseases center, Beijing Ditan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTH-XY002
Record Dates: First submitted 2011-10-31; First posted 2011-11-15 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peginterferon alpha 2a (Experimental): the inactive chronic HBsAg carriers were treated with peginterferon alpha 2a for 72 weeks and followed for 24 weeks.
  Interventions: Drug: Pegylated interferon alfa-2a

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a — patients were given peginterferon alfa-2a (40KD) (Pegasys®; Roche, Basel, Switzerland)180 µg by subcutaneous injection once weekly for 120 weeks
  Other Names: Pegasys®; Roche, Basel, Switzerland

SUMMARY:
Hepatitis B surface antigen loss/seroconversion, considered to be the ideal outcome of chronic hepatitis B virus (HBV) infection, occurs spontaneously at a low rate in inactive carriers.

The researchers aim to investigate the ability of peginterferon alpha-2a to achieve surface antigen loss/seroconversion therapy in inactive carriers with persistently normal alanine aminotransferase (ALT) levels, undetectable HBV DNA and low surface antigen levels, who would not generally be considered candidates for therapy.

DETAILED DESCRIPTION:
Chronic HBV inactive carriers were enrolled in the out-patient department of Beijing Ditan Hospital. All of them were HBsAg positive and anti-HBs negative for more than 6 months with persistent undetectable HBV DNA and normal ALT levels measured at 3-6 monthly intervals during the preceding 2 years as well as with serum HBsAg levels ≤100 IU/mL determined on two occasions during the month prior to treatment. All patients did not have other liver diseases and contraindications for interferon therapy.

After giving informed consent, patients were treated with weekly subcutaneous injections of peginterferon alpha-2a 180 µg. The use of other immune suppressive or regulatory drugs and other antiviral drugs was prohibited during the course of the study.

In this study, the only parameter to assessing the treatment response was HBsAg level change. Treatment endpoint was HBsAg loss(<0.05 IU/mL) and anti-HBs positive(>10 mIU/mL) defined as seroconversion.

Depending on the decline of HBsAg level, treatment was either continued for a prolonged period until the endpoint was achieved, or terminated in case of nonresponse. Treatment was proceeded if HBsAg level continued to decline until HBsAg seroconversion was achieved and the anti-HBs level was above 200 mIU/ml. If the patients were not willing to extend treatment, the therapy was ended at the time of HBsAg loss, or stopped without further decline of HBsAg levels on three months treatment.

Liver function parameters, including ALT, aspartate aminotransferase (AST), albumin (ALB) and total bilirubin (Tbil) were examined using an automated biochemical analyzer. Peripheral blood neutrophil and platelet count were detected before treatment, and monitored during treatment with one to three month intervals, and base on the test results to adjust the next checking time. Quantitative HBV DNA testing was conducted using a commercially available real-time fluorescence quantitative PCR kit. HBsAg levels were quantified with Architect i2000 HBsAg quantitative assay (Abbott Laboratories) kit.

The main efficacy endpoints were HBsAg loss and seroconversion.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive and anti-HBs negative for more than 6 months
* HBeAg-negative/anti-HBe-positive
* Persistently undetectable HBV DNA with normal ALT levels, as established at 3-6 monthly intervals during the preceding 2 yrs
* Serum HBsAg levels ≤100 IU/mL, as determined on two occasions during the month prior to treatment
* Absence of previous antiviral therapy

Exclusion Criteria:

* With active alcohol and/or drugs consumption
* With human immunodeficiency virus or hepatitis C virus coinfections
* With clinical evidence of cirrhosis
* With history of autoimmune hepatitis
* With hematological or psychiatric diseases
* With evidence of neoplastic diseases
* With severe cardiac or pulmonary disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HBsAg loss/seroconversion | HBsAg level was lower than 0.05IU/mL after 96 weeks treatment
  HBsAg loss was defined as HBsAg levels <0.05 IU/mL. Anti-HBs was measured using Architect i2000 kit,and anti-HBs >10 mIU/L was considered positive.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, phD/MD, Principal Investigator — Liver diseases center, Beijing Ditan Hospital
Locations (1):
- liver disease center, Beijing Ditan Hospital, Beijing, Beijing Municipality, China